CLINICAL TRIAL: NCT00346567
Title: Clinical Trial: Backup With Combivir (AZT/3TC) or Single Dose (sd) Truvada (FTC/TDF) in Order to Avoid NNRTI Resistance After sd Nevirapine for the Prevention of Mother-to-child Transmission (MTCT)
Brief Title: Backup With Combivir or Single Dose (SD) Truvada in Order to Avoid Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) Resistance After SD Nevirapine for the Prevention of Mother-to-child Transmission (PMTCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Terese Katzenstein Consultant, MD, Ph.D. DMSc, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: comtru
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: mother-to-child-transmission; PMTCT; HIV; resistance; NNRTI
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Lamivudine; lamivudine, zidovudine drug combination; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

ARMS (2):
- 1 (Active Comparator): AZT from week 28 or asap thereafter. Intrapartum AZT and 3TC + Single dose NVP Postpartum Combivir tail for 7 days twice daily
  Interventions: Drug: Zidovudine and Lamivudine (Combivir)
- 2 (Experimental): AZT from week 28 or asap thereafter. Intrapartum Single dose Truvada + Single dose NVP
  Interventions: Drug: Emtricitabine and Tenofovir (Truvada)

INTERVENTIONS:
Drug: Zidovudine and Lamivudine (Combivir)
  Arms: 1
Drug: Emtricitabine and Tenofovir (Truvada)
  Arms: 2

SUMMARY:
The aim of the study is to find short course alternatives to single dose (sd)nevirapine for the prevention of mother-to-child HIV-transmission with the same or better degree of transmission protection than sd nevirapine but with less NNRTI resistance development.

DETAILED DESCRIPTION:
Randomised open study comparing Zidovudine from 28 weeks gestation, single dose Nevirapine + 1 week of Combivir with Zidovudine from 28 weeks gestation, single dose Nevirapine + single dose of Truvada for the mothers during birth. In both arms the infants will receive one dose of nevirapine within the first days after births as well as 7 to 28 days Zidovudine. N = 450. The study will be conducted at Ngamiani and Makorora Health Centres and Bombo Regional Hospital in Tanga, Tanzania as a cooperation between Rigshospitalet, Denmark, University of Copenhagen and National Institute of Medical Research, Tanzania.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected, antiretroviral naive, not fulfilling national Tanzanian criteria for HAART treatment, giving informed consent, consenting to homevisit-follow-up in case of no-show for scheduled hospital visit.

Exclusion Criteria:

* CD4 less than 350 x10(6)/L, suffering from systemic diseases in need of medical treatment e.g. TB, renal or liver failure etc.
* Creatinin higher than 1,5 mg/dL, Alanine aminotransferase above 140 U/L

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 566 (Actual)
Dates: Start 2006-06; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
frequency of mother-to-child HIV transmission | 6 weeks post partum
frequency of NNRTI resistance development | 6 weeks post partum

SECONDARY OUTCOMES:
Comparison of p24 antigen to HIV RNA for treatment induced changes in viremia | Delivery, day 7, day 42 and month 9 post partum
Comparison of p24 antigen ability to detect viremia for the various subtypes A,C & D | Delivery, Day 7, Day 42 post partum, mother, Day 42 and Day 90 post partum child

CONTACTS AND LOCATIONS:
Overall Officials: Terese L Katzenstein, MD Ph.D., Study Director — Rigshospitalet, Denmark
Locations (1):
- Bombo Regional Hospital, Tanga, Tanzania